CLINICAL TRIAL: NCT05431595
Title: Managing Agitated Delirium With Neuroleptics and Anti-Epileptics as a Neuroleptic Sparing Strategy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0172; NCI-2022-05252 (Other: NCI-CTRP Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Delirium; Epileptics; Neuroleptics
MeSH Terms: conditions — Delirium; Epilepsy | interventions — Haloperidol; Chlorpromazine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Participants will receive haloperidol by vein every 12 hours (or more often, as needed).
  Interventions: Drug: Haloperidol
- Group 2 (Experimental): Participants will receive chlorpromazine by vein every 12 hours (or more often, as needed).
  Interventions: Drug: Chlorpromazine
- Group 3 (Experimental): Participants will receive valproate by vein every 12 hours.
  Interventions: Drug: Valproate
- Group 4 (Experimental): Participants will receive placebo every by vein every 12 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — Given by Vein (IV)
  Arms: Group 1
Drug: Chlorpromazine — Given by Vein (IV)
  Other Names: Chlorpromazine hydrochloride, Thorazine®
  Arms: Group 2
Drug: Valproate — Given by Vein (IV)
  Other Names: Depakene; Valproate Acid
  Arms: Group 3
Drug: Placebo — Given by Vein (IV)
  Arms: Group 4

SUMMARY:
To examine the effects of haloperidol, chlorpromazine, valproic acid and placebo, in conjunction with standardized non-pharmacologic interventions, in the first line treatment of agitated delirium in hospitalized patients with cancer. This double-blind, randomized clinical trial aims to provide evidence on various therapeutic options for palliating delirium, thereby reducing delirium-related distress and ultimately alleviating suffering.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

Compare the effect of scheduled haloperidol, chlorpromazine, valproate and placebo (non-pharmacological interventions alone) on the frequency of breakthrough restlessness over 72 hours in patients with agitated delirium seen by the palliative care consultation team. Our working hypothesis is that haloperidol, chlorpromazine, and valproate will lead to fewer episodes of breakthrough restlessness than placebo.

Secondary Objective #1:

Compare the effects of scheduled haloperidol, chlorpromazine, valproate and placebo on (1) RASS-PAL, (2) need for dose escalation, (3) perceived comfort by caregivers and bedside nurses, (4) delirium severity (Memorial Delirium Assessment Scale), (5) delirium-related distress in caregivers and nurses (Delirium Experience Questionnaire), (6) delirium recall in patients (Delirium Recall Questionnaire), (7) symptom expression (Edmonton Symptom Assessment Scale), (8) adverse effects, and (9) survival. Our working hypothesis is that haloperidol, chlorpromazine, and valproate are superior to placebo (non-pharmacologic interventions alone) in improving delirium-related outcomes.

Secondary Objective #2:

Estimate the efficacy of non-pharmacologic interventions alone on breakthrough restlessness. Our working hypothesis is that patients in the placebo group will require fewer breakthrough doses in the 72 hours after implementation of non-pharmacological interventions

ELIGIBILITY:
Inclusion Criteria:

1. [Patients] Diagnosis of advanced cancer (defined as locally advanced, metastatic recurrent, or incurable disease)
2. [Patients] Seen by palliative care inpatient consultation team
3. [Patients] Delirium as per DSM-5 criteria
4. [Patients] Hyperactive or mixed delirium with either a rescue medication order or any non-pharmacologic measures (e.g. sitter, restraints) for agitation, restlessness, or delirium
5. [Patients] Age 18 years or older
6. [Patients] Permission from clinician from primary team to enroll
7. [Family Caregivers] Patient's spouse, adult child, sibling, parent, other relative, or significant other (defined by the patient as a partner)
8. [Family Caregivers] Age 18 years or older

Exclusion Criteria:

1. [Patients] On scheduled haloperidol >4 mg/d, chlorpromazine >100 mg/d, or valproate >750 mg/d
2. [Patients] History of myasthenia gravis, acute narrow-angle glaucoma, or hepatic encephalopathy as documented in chart
3. [Patients] Hepatic dysfunction (unresolved AST or ALT >2.5x ULN, bilirubin >1.5x ULN or INR >1.5 within past month)
4. [Patients] History of neuroleptic malignant syndrome as documented in chart
5. [Patients] Active seizure disorder within past month as documented in chart
6. [Patients] History of Parkinson's disease or dementia as documented in chart
7. [Patients] History of prolonged QTc interval (>500 ms) if documented by most recent ECG within the past month
8. [Patients] Hypersensitivity to haloperidol, chlorpromazine, or valproate as documented in chart
9. [Patients] Pancreatitis within past month as documented in chart
10. [Patients] Currently on lamotrigine, phenobarbital, or carbamazepine
11. [Patients] Physical signs of impending death such as respiration with mandibular movement and death rattle
12. [Patients] Pregnancy as documented in chart
13. [Patients] Active COVID-19 infection as documented in chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment Scale Questionnaire | through study completion, an average of 1 year
  Edmonton Symptom Assessment Scale (ESAS)-score scale ranges from (0-10) No pain-0/Worse Possible Pain 10 (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org